CLINICAL TRIAL: NCT04325503
Title: Neurobiological Drivers of Mobility Resilience: The Dopaminergic System
Acronym: RES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00156490; 5U01AG061393-05 (NIH)
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Parkinsonian Signs in Older Persons
Keywords: slow gait; Parkinsonian signs
MeSH Terms: interventions — Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): carbidopa and carbidopa-levodopa treatment for parkinsonian signs in older persons using standard dosing, frequency for a duration for 1-2 weeks
  Interventions: Drug: carbidopa

INTERVENTIONS:
Drug: carbidopa — carbidopa and carbidopa-levodopa standard treatment
  Other Names: carbidopa-levodopa

SUMMARY:
Walking with age becomes both slower and less 'automated', requiring more attention and brain resources. As a result, older adults have a greater risk of negative outcomes and falls. There is an urgent need to identify factors that can help compensate for these harmful factors and reduce walking impairments, as there are currently no effective treatments available. Investigators have recently discovered that ~20% of older adults maintain fast walking speed even in the presence of small blood vessel brain changes and leg problems, thus appearing to be protected against these harmful factors. The investigators work suggests that the brain dopamine (DA) system may be a source of this protective capacity. Investigators have also shown that lower levels of dopamine are associated with slow walking. Investigators will be investigating the role of dopamine on slow walking and other parkinsonian signs using detailed clinical assessment, assessment of dopamine activity, and clinical interventions.

DETAILED DESCRIPTION:
Walking with age becomes both slower and less 'automated', requiring more attention and prefrontal resources. As a result older adults have a greater risk of adverse mobility outcomes and falls. Walking disturbances in the elderly have been linked to changes in both cerebral, in particular small vessel disease (cSVD), and peripheral systems. There is an urgent need to identify factors that can help compensate for these harmful factors and reduce walking impairments, as there are currently no effective treatments available. Although effective mobility is the end result of the functional capacity of both central and peripheral systems, the brain's unique modulatory and adaptive capacity may provide clues for novel interventions. For example, investigators have recently discovered that ~20% of older adults maintain fast walking speed even in the presence of age related cSVD and peripheral system impairments, thus appearing resilient to these harmful factors. The investigators work suggests that the nigrostriatal dopamine (DA) system may be a source of this resilience. As investigators recent findings suggest, DA neurotransmission positively predicts walking speed; it also attenuates the negative effects of age related cSVD and peripheral system impairments on walking speed. These findings are consistent with post-mortem evidence that a combination of loss of nigral DA neurons and cSVD best predict age-related walking impairment. The nigrostriatal DA system plays a critical role in motor control; nigrostriatal. DA neurotransmission regulates the automated execution of overlearned motor tasks via its connections with sensorimotor cortical and subcortical areas.

The investigators hypothesize that higher nigrostriatal DA neurotransmission drives resilience to cSVD and peripheral system impairments, via higher connectivity of sensorimotor networks, thus increasing automaticity of walking and reducing prefrontal engagement while walking. Unlike cSVD and brain structural impairments, DA neurotransmission is potentially modifiable, thereby offering novel approaches to treat non-resilient elderly in a targeted fashion. This translational pilot study will use a biomechanistic target engagement study in older adults with slow walking and/or other parkinsonian signs.

The study will include elderly men and women age 60 or older with evidence of mild parkinsonian signs (MPS, or slow gait (< 1m/s)) and/or additional cSVD on brain MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 or older (M/F)
2. Evidence of mild parkinsonian signs (incl. slow gait (< 1m/s))

Exclusion Criteria:

1. Presence of clinically significant degenerative joint disease and/or neuropathy interfering with proper assessment of the motor UPDRS exam.
2. Presence of significant dementia.
3. Evidence of a large vessel stroke in a clinically relevant area (cerebral cortex, basal ganglia, thalamus) or mass lesion on structural brain imaging (MRI).
4. Participants in whom magnetic resonance imaging (MRI) is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant.
5. Severe claustrophobia precluding neuroimaging procedures.
6. Hypersensitivity to the carbidopa, levodopa, and tablet components.
7. Any other medical history determined by investigators to preclude safe participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Bohnen, MD, Principal Investigator — University of Michigan
Locations (1):
- Functional Neuroimaging, Cognitive, and Mobility Lab, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Results will be provided in publications

RESULTS

PARTICIPANT FLOW:
Groups:
- Carbidopa and Carbidopa-Levodopa Treatment: All participants treated with 25 mg carbidopa three times daily (TID) and 1.5 pills of 25/100 mg carbidopa-levodopa TID for parkinsonian signs in older persons (standard dosing, frequency for a duration for 1-2 weeks).
Period: Overall Study
Arm/Group | Carbidopa and Carbidopa-Levodopa Treatment
Started | 14
Completed | 11
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — PI decided to remove them from trial as they lacked motor symptoms being studied. | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (6.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Average Gait Speed [Mean (Standard Deviation); unit: meters/second] — Average gait speed as measured using wearable sensors worn during walking tasks. Gait speed is measured in meters per second. Population: Average gait speed was not collected for 3 participants because they withdrew (Two participants were withdrawn from the study due to lack of motor symptoms. One participant withdrew from study due to personal time constraints). Gait data was not collected for one participant due to software error.
  meters/second
    number analyzed (Participants) | 10
    (all) | 0.882 (0.072)
Montreal Cognitive Assessment (MoCA) Score [Mean (Standard Deviation); unit: score on a scale] — Cognitive assessment used to evaluate individuals for mild cognitive impairment. Scores range from 0-30. Higher scores indicate better performance. Population: MoCA was not collected for 3 participants because they withdrew from the study (two participants were withdrawn from the study due to lack of motor symptoms. One participant withdrew from study due to personal time constraints).
  score on a scale
    number analyzed (Participants) | 11
    (all) | 26.27 (2.76)
Mini Balance Evaluation Systems Test (Mini-BESTest) [Mean (Standard Deviation); unit: score on a scale] — The mini-BESTest is a 14-item evaluation of dynamic balance and postural control. It is scored from 0-28, with higher scores indicating better performance. Population: Mini-BESTest was not collected for 3 participants because they withdrew from the study (two participants were withdrawn from the study due to lack of motor symptoms. One participant withdrew from study due to personal time constraints).
  score on a scale
    number analyzed (Participants) | 11
    (all) | 20.09 (4.253)
Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III total [Mean (Standard Deviation); unit: units on a scale] — MDS-UPDRS part III is the motor examination portion of the UPDRS evaluation. Scores range from 0-132, with higher scores indicating greater severity of motor symptoms.
  units on a scale | 29.93 (11.672)
Short Activities-specific Balance Confidence (sABC) scale score [Median (Full Range); unit: score on a scale] — Participants rate their level of confidence in doing specific activities without losing their balance as a percentage, with 0% indicating they are certain they would lose their balance and 100% indicating that they are certain they can complete the task without losing their balance. Scores on these 6 questions are averaged to determine total sABC score. Scores range from 0-100, with higher scores indicating greater balance confidence. Population: sABC was not collected for 3 participants because they withdrew from the study (two participants were withdrawn from the study due to lack of motor symptoms. One participant withdrew from study due to personal time constraints). One participant did not complete questionnaire due to tech error.
  score on a scale
    number analyzed (Participants) | 10
    (all) | 76.67 [23.33 to 95.00]
Cognitive z-score [Mean (Standard Deviation); unit: Z-score] — Composite variable calculated based on the Stroop Color Word Interference test I-IV (assessment of attention) and Delis-Kaplan Executive Function System Trail Making test I-V (assessment of executive function and working memory), adjusted based on normative data for older adults. A z-score of 0 represents the control population mean. Scores above the mean indicate better performance, while scores below the mean indicate poorer performance. Population: Cognitive z-scores were not collected for 3 participants because they withdrew from the study (two participants were withdrawn from the study due to lack of motor symptoms. One participant withdrew from study due to personal time constraints). One participant did not complete all cognitive testing due to language barrier.
  Z-score
    number analyzed (Participants) | 10
    (all) | -0.151 (0.751)
Wechsler Adult Intelligence Scale Digit Symbol Test Score [Mean (Standard Deviation); unit: score on a scale] — Evaluation of cognitive functioning in which a participant is given a key of numbers 1-9, each paired with a unique symbol. Below the key, is a series of random numbers which they participant must fill in the corresponding symbol for. They have 120 seconds to complete the task. Participants receive one point for each correct symbol written. Score range from 0-133. Population: The digit symbol test was not collected for 3 participants because they withdrew from the study (two participants were withdrawn from the study due to lack of motor symptoms. One participant withdrew from study due to personal time constraints). Two participants did not complete testing due to tech error.
  score on a scale
    number analyzed (Participants) | 9
    (all) | 54.67 (22.472)

OUTCOME MEASURES:

1. Primary Outcome: Average Gait Speed
Description: Average gait speed as measured using wearable sensors worn during walking tasks. Gait speed is measured in meters per second.
Time Frame: 7-13 days after beginning treatment.
Population: Gait speed data was missing for one participant due to software error.
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Carbidopa and Carbidopa-Levodopa Treatment
Number analyzed (Participants) | 10
meters/second | 0.973 (0.123)
Statistical Analysis 1: Comparison: Carbidopa and Carbidopa-Levodopa Treatment; Test type: Other — A comparison is not being made between two different treatment groups; p = 0.015, t-test, 2 sided — A priori threshold statistical significance p < 0.05; Paired samples t-test, df = 9; Mean Difference (Net) = 0.0905, 95% CI 2-sided [0.022 to 0.159]

2. Primary Outcome: Montreal Cognitive Assessment (MoCA)
Description: Cognitive assessment used to evaluate individuals for mild cognitive impairment. Scores range from 0-30. Higher scores indicate better performance.
Time Frame: 7-13 days after beginning treatment
Population: Two participants did not complete the MoCA during the follow-up visit due to time constraints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carbidopa and Carbidopa-Levodopa Treatment
Number analyzed (Participants) | 9
score on a scale | 27.44 (1.59)
Statistical Analysis 1: Comparison: Carbidopa and Carbidopa-Levodopa Treatment; Test type: Other — A comparison is not being made between two different treatment groups; p = 0.694, t-test, 2 sided — A priori threshold for statistical significance is p < 0.05; Paired samples t-test, df = 8; Mean Difference (Net) = 0.333, 95% CI 2-sided [-1.550 to 2.216]

3. Primary Outcome: Mini Balance Evaluation Systems Test (Mini-BESTest)
Description: The mini-BESTest is a 14-item evaluation of dynamic balance and postural control. It is scored from 0-28, with higher scores indicating better performance.
Time Frame: 7-13 days after beginning treatment
Population: Testing was not completed for two participants due to time constraints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carbidopa and Carbidopa-Levodopa Treatment
Number analyzed (Participants) | 9
score on a scale | 22.89 (3.951)
Statistical Analysis 1: Comparison: Carbidopa and Carbidopa-Levodopa Treatment; Test type: Other — A comparison is not being made between two different treatment groups; p = 0.103, t-test, 2 sided — A priori threshold for statistical significance was p < 0.05; Paired samples t-test, df = 8; Mean Difference (Net) = 1.444, 95% CI 2-sided [-0.363 to 3.252]

4. Primary Outcome: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III Total
Description: MDS-UPDRS part III is the motor examination portion of the UPDRS evaluation. Scores range from 0-132, with higher scores indicating greater severity of motor symptoms.
Time Frame: 7-13 days after beginning treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Carbidopa and Carbidopa-Levodopa Treatment
Number analyzed (Participants) | 11
units on a scale | 31.18 (10.998)
Statistical Analysis 1: Comparison: Carbidopa and Carbidopa-Levodopa Treatment; Test type: Other — A comparison is not being made between two different treatment groups; p = 0.321, t-test, 2 sided — A priori threshold for statistical significance p < 0.05; Paired samples t-test, df = 10; Mean Difference (Net) = -2.09, 95% CI 2-sided [-6.554 to 2.372]

5. Primary Outcome: Cognitive Z-score
Description: Composite variable calculated based on the Stroop Color Word Interference test I-IV (assessment of attention) and Delis-Kaplan Executive Function System Trail Making test I-V (assessment of executive function and working memory), adjusted based on normative data for older adults. A z-score of 0 represents the control population mean. Scores above the mean indicate better performance, while scores below the mean indicate poorer performance.
Time Frame: 7-13 days after beginning treatment
Population: Data was not collected for 3 participants (one participant did not complete Stroop Color Word Interference tests due to language barrier. One participant did not complete cognitive assessments due to poor vision interfering with test-taking ability. One participant did not complete cognitive testing due to time constraints).
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Carbidopa and Carbidopa-Levodopa Treatment
Number analyzed (Participants) | 8
Z-score | 0.271 (0.524)
Statistical Analysis 1: Comparison: Carbidopa and Carbidopa-Levodopa Treatment; Test type: Other — A comparison is not being made between two different treatment groups; p = 0.265, t-test, 2 sided; Paired samples t-test, df = 7; Mean Difference (Net) = 0.185, 95% CI 2-sided [-0.175 to 0.544]

6. Primary Outcome: Wechsler Adult Intelligence System Digit Symbol Substitution Test
Description: Evaluation of cognitive functioning in which a participant is given a key of numbers 1-9, each paired with a unique symbol. Below the key, is a series of random numbers which they participant must fill in the corresponding symbol for. They have 120 seconds to complete the task. Participants receive one point for each correct symbol written. Score range from 0-133.
Time Frame: 7-13 days after beginning treatment
Population: Two participants did not complete testing due to time constraints
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carbidopa and Carbidopa-Levodopa Treatment
Number analyzed (Participants) | 9
score on a scale | 65.89 (20.829)
Statistical Analysis 1: Comparison: Carbidopa and Carbidopa-Levodopa Treatment; Test type: Other — A comparison is not being made between two different treatment groups; p = 0.0270, t-test, 2 sided — A priori threshold for statistical significance p < 0.05; Paired samples t-test, df = 6; Mean Difference (Net) = 8.143, 95% CI 2-sided [1.296 to 15.0]

7. Secondary Outcome: Short Activities-specific Balance Confidence Scale Score
Description: Participants rate their level of confidence in doing specific activities without losing their balance as a percentage, with 0% indicating they are certain they would lose their balance and 100% indicating that they are certain they can complete the task without losing their balance. Scores on these 6 questions are averaged to determine total sABC score. Scores range from 0-100, with higher scores indicating greater balance confidence.
Time Frame: 7-13 days after beginning treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Carbidopa and Carbidopa-Levodopa Treatment
Number analyzed (Participants) | 11
score on a scale | 70.00 [21.67 to 93.3]
Statistical Analysis 1: Comparison: Carbidopa and Carbidopa-Levodopa Treatment; Test type: Other — A comparison is not being made between two different treatment groups; p = 0.153, Wilcoxon (Mann-Whitney) — A priori threshold for statistical significance p < 0.05

ADVERSE EVENTS:
Time Frame: Up to 14 days
Arm/Group | Carbidopa and Carbidopa-Levodopa Treatment
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 8/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbidopa and Carbidopa-Levodopa Treatment (N=14)
Nausea (Gastrointestinal disorders) | 4 (4) — Mild, expected Adverse event (AE).
Vivid dreams (General disorders) | 2 (2) — Mild, expected AE.
Mild Changes to Bowel Movement (Gastrointestinal disorders) | 1 (1) — Mild, expected AE.
Mild Nasal Congestion (General disorders) | 2 (2) — Mild, unexpected AE.
Anxiety (Psychiatric disorders) | 1 (2) — Mild, expected AE.
Headache (General disorders) | 2 (2) — Mild, expected AE.
Change in Blood Glucose Level (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT04325503/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT04325503/ICF_000.pdf